CLINICAL TRIAL: NCT00333827
Title: Multicenter Randomized Study Of Cell Therapy In Cardiopathies - Dilated Cardiomyopathy
Brief Title: Cell Therapy In Dilated Cardiomyopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Bernardo Rangel Tura, Professor, Ministry of Health, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMRTCC-MCD
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Dilated Cardiomyopathy
Keywords: Dilated Cardiomyopathy; stem cells; Therapeutics; Randomized Controlled Trials
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Carboxylesterase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Optimal Therapy (Active Comparator): Optimal therapy for cardiac failure
  Interventions: Drug: optimal therapy for cardiaca failure
- cell therapy (Experimental): stem cell
  Interventions: Procedure: cell

INTERVENTIONS:
Drug: optimal therapy for cardiaca failure — optimal therapy for cardiaca failure
  Arms: Optimal Therapy
Procedure: cell — stem cell
  Arms: cell therapy

SUMMARY:
The purpose of this study is to determine effect of cell therapy in patients with severe dilated cardiomyopathy

DETAILED DESCRIPTION:
This protocol describes a double-blind placebo controlled randomized clinical trial to evaluate the efficacy of bone marrow derived stem cell implants in 300 bazillion patients with dilated cardiomyopathy and heart failure in class III or IV of the New York Heart Association.

The primary endpoint of this study is to evaluate the effect of the autologous bone marrow stem cell implant in the increase of the ejection fraction of the left ventricle in comparison with a control group, under optimized therapy for dilated cardiomyopathy. Secondary endpoints will evaluate the alteration in NYHA functional class, mortality rate, physical capacity (by ergoespirometry), life quality (Minnesota questionnaire) and pulmonary congestion in dilated cardiomyopathy patients the received the autologous bone-marrow stem cell implant.

Hypothesis: The main hypothesis of this study is that the patients who received the autologous bone-marrow stem cell implant will have after a 6 month follow-up a mean 5% increase in absolute left ventricle ejection fraction in comparison with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dilated cardiomyopathy according to WHO criteria
* Syndromic heart failure in functional class III or IV of the NYHA
* Enrollment and continuous follow-up in cardiac out-patient clinic
* Adequate medical therapy after optimization therapy
* Echocardiogram with an ejection fraction equal to or less than 35% by Simpson's rule

Exclusion Criteria:

* Valvular diseases, except functional mitral or tricuspid reflow
* Coronariography showing a significant lesion (obstruction of at least 50% of the lumen in the troncus or the main arteries - LAD, CX, RC) in one or more arteries
* Serologic diagnosis for Chagas disease or at least two of the following criteria: epidemiology, right bundle branch block, anterior hemi-block, apical aneurism
* Sustained ventricular tachycardia
* Abusive use of alcohol or illicit drugs
* Pregnancy
* Use of cardio toxic drugs
* Any co-morbidity with impact in life expectancy in 2 years
* Renal function compromised (creatinine above 2 mg/dl)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
increase of the ejection fraction of the left ventricle | 6 months

SECONDARY OUTCOMES:
Death by any cause | 1 year
Maximum oxygen consumption difference, as measured by ergoespirometry, at six and twelve months in relation to baseline | 1 year
Difference in life quality as estimated by Minnesota living with Heart Failure Questionnaire | 6 month
Difference in NYHA functional class | 6 month
Percent number of patients that reached an absolute increase of 5% in ejection fraction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carlos C de Carvalho, MD,PhD, Study Director — INCL; Bernardo R Tura, Md,MsC, Study Chair — INCL; Augusto Z Bozza, MD, Principal Investigator — INCL
Locations (1):
- INCL - National Institute of Cardiology Laranjeiras, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Martino H, Brofman P, Greco O, Bueno R, Bodanese L, Clausell N, Maldonado JA, Mill J, Braile D, Moraes J Jr, Silva S, Bozza A, Santos B, Campos de Carvalho A; Dilated Cardiomyopathy Arm of the MiHeart Study Investigators. Multicentre, randomized, double-blind trial of intracoronary autologous mononuclear bone marrow cell injection in non-ischaemic dilated cardiomyopathy (the dilated cardiomyopathy arm of the MiHeart study). Eur Heart J. 2015 Nov 7;36(42):2898-904. doi: 10.1093/eurheartj/ehv477. Epub 2015 Sep 20. PMID 26392433